CLINICAL TRIAL: NCT03031600
Title: Pilot Validation of a Hemodilution Technique to Estimate Blood Volume in Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Duke University (Other); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: HU0001-16-1-TS14(N16-P10)
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Hypovolemia; Hypervolemia
MeSH Terms: conditions — Hypovolemia; Edema

STUDY DESIGN:
Intervention Model Description: This study will use a prospective validation design. In this design, each subject will experience both estimation methods/arms (radiodilution and hematocrit dilution) in a fixed sequence. The fixed order is necessary, as hematocrit dilution would bias the results of radiodilution by iatrogenically increasing plasma volume as part of the estimation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiodilution via Daxor BVA-100 (Active Comparator): In study arm 1, actual blood volume will be measured using the Daxor Blood Volume Analyzer-100 (BVA-100). In this technique, the subject is injected with 1 ml of human serum albumin labeled with iodine131 (25 microcuries). A small amount of blood is collected from the subject just before injection and at 12, 18, 24, 30, and 36 min after injection.
  Interventions: Diagnostic Test: Radiodilution via Daxor BVA-100
- Hemodilution via hematocrit measurement (Experimental): In study arm 2, estimated blood volume will measured via hemodilution. . A blood sample (5 ml) will be drawn for baseline determination of hematocrit via iSTAT and lab measurement from the non-dominant arm. After the baseline hematocrit blood sample is drawn, a volume of normal saline equivalent to 10% of the subject's ideal blood volume will be administered over a 12-minute period through the dominant arm IV catheter. Twelve minutes after the infusion is complete, a second blood sample (5 ml) will be drawn from the non-dominant arm for determination of post-bolus hematocrit via iSTAT and lab. Subjects will then be asked to void into a urinal, and urine output will be measured in ml.
  Interventions: Diagnostic Test: Hemodilution via hematocrit measurement

INTERVENTIONS:
Diagnostic Test: Radiodilution via Daxor BVA-100 — The BVA-100 measures the hematocrit and residual plasma radioactivity of each sample in a semi-automated process, and the residual radioactivity is compared from that of the pre-injection sample to determine plasma volume. The plasma volume and BVA-100-measured hematocrit are then used to calculate the red cell volume and actual blood volume. The BVA-100 is FDA approved for blood volume measurement in vivo, has a reported precision of ± 2.5%, and has demonstrated accuracy and specificity in blood volume assessment in clinical and research settings (Van, P.Y., et al., 2011, Borovka, M., et al., 2013).
  Arms: Radiodilution via Daxor BVA-100
Diagnostic Test: Hemodilution via hematocrit measurement — Hemodilution uses the ideal blood volume and serial hematocrit measures drawn before and after administration of a known quantity of IV fluid to estimate blood volume. Ideal blood volume is calculated using the methods described by Feldschuh and colleagues (Feldschuh, J. and Y. Enson, 1977; Feldschuh, J. and S. Katz, 2007). Hematocrit is measured using the Abbot iSTAT point of care testing device and the lab. Urine output is measured in ml. The ideal blood volume, pre and post-bolus hematocrit, fluid bolus volume, and urine output will be used to calculate estimated blood volume using a mathematical model previously described by the investigators (D'Angelo, M., et al., 2015).
  Arms: Hemodilution via hematocrit measurement

SUMMARY:
The objective of this study is to determine the accuracy of estimating patient blood volume using field-expedient point-of-care measurement of hematocrit before and after hemodilution with a standardized volume of intravenous solution, in comparison to determining patient blood volume by radiodilution. A total of 33 healthy adult male subjects aged 18-35 years will undergo determination of blood volume in a fixed order: first by radiodilution, then by hemodilution. Blood volume as measured by radiodilution will be correlated with blood volume as estimated with hemodilution to assess the potential validity of hemodilution as means of estimating blood volume.

DETAILED DESCRIPTION:
The primary goal of perioperative fluid therapy is to optimize patient blood volume for a given degree of cardiac function and thereby promote adequate end organ tissue perfusion. In the ideal situation, a surgical patient would maintain a euvolemic total blood volume (TBV) that promotes optimal tissue oxygenation, nutrient supply, and removal of metabolic waste products. Current methods to assess perioperative TBV and manage intravenous (IV) fluids, which include fluid algorithms, physiologic parameters, blood studies, and clinician intuition, are either inaccurate or require highly specialized equipment and training. Therefore, clinicians are faced with the formidable task of attempting to titrate IV fluids with the goal of preserving optimal tissue perfusion in the perioperative period without knowledge of the patient's actual TBV. This long standing clinical conundrum, and the potential iatrogenic consequences of hypo- or hypervolemia, has recently produced a significant degree of inquiry into direct and indirect methods to evaluate cardiac output as a product of fluctuating TBV. The goal of much of this investigation is to generate an evidence-based methodology for administration of perioperative IV fluids to promote euvolemia and preserve adequate tissue perfusion. There is strong evidence from the civilian anesthesia and surgical literature that the use of various indicators of cardiac output as a marker of TBV and a guide for fluid therapy, so called Goal Directed Fluid Therapy (GDFT), leads to significantly better perioperative patient outcomes. However, current GDFT management protocols rely heavily on technology not readily available within or sufficiently ruggedized for use in the military field setting where ongoing accurate estimation of TBV to guide fluid replacement in the presence of major trauma, and its physiologic aftermath, may be critical to survival. Therefore, the primary objective of this study is to assess the accuracy of determining patient TBV using measurement of red blood cell volume (hematocrit, or HCT) with a point-of-care testing device relevant to the military setting, before and after hemodilution with a standard IV solution. The specific aims of the proposed research are to:

1. Determine subject total blood volume using the gold standard DAXOR Blood Volume Analyzer-100 Analysis System (Radiotracer Dilution Technique).
2. Compute estimated subject total blood volume using venous blood hematocrit values drawn before and after an intravenous fluid bolus (Hemodilution Technique).
3. Correlate inter-subject radiotracer dilution technique-derived total blood volume with hemodilution technique-derived total blood volume.

Hypothesis:

The calculated total blood volume derived by a simple clinically applicable hemodilution technique will highly correlate with the gold standard laboratory radiotracer dilution technique.

The proposed study will examine the utility of a simple, clinically applicable, and adaptable method to assess a patient's TBV that does not rely on sophisticated, technology-dependent, direct or indirect measures of cardiac output. Development and confirmation of the accuracy of a simple method to intermittently determine a patient's TBV in the perioperative setting would revolutionize the ability of a practitioner to match perioperative IV fluid administration to the goal of optimizing cardiac output and tissue perfusion. The tremendous potential positive impact of this work on surgical and anesthesia care in both the military and civilian settings is evident in the brief but expansive existing work demonstrating significant improvement in patient outcomes using GDFT techniques. The proposed study is potentially the first step in a future program of research to bring the benefits of GDFT into austere settings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal body mass index (defined as 18.5-24.9 per guidelines issued by the Centers for Disease Control and Prevention)

Exclusion Criteria:

* Otherwise eligible subjects one or more of the following conditions will be excluded from participation due to the potential to alter blood volume, plasma volume, red cell volume, or microvascular circulation: Cardiovascular disease (to include hypertension, congestive heart failure, previous myocardial infarction, valvular heart disease other than asymptomatic mitral valve prolapse, cardiomyopathy, or peripheral vascular disease), endocrine disease (to include syndrome of inappropriate diuretic hormone, diabetes insipidus, hypothyroidism, hyperthyroidism, or diabetes mellitus), adrenal insufficiency or hypersecretion, renal failure or insufficiency, liver disease, history of sepsis, intravenous fluid administration, nausea, vomiting, diarrhea or heat stress injury within 30 days of the test, eating disorders such as bulimia or anorexia nervosa, or current diuretic or antihypertensive medication use.
* Additionally, subjects who are allergic to iodine, albumin, or iodinated I131 albumin, or cannot undergo intravenous catheter placement will be ineligible to participate.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between actual and estimated blood volume | Actual blood volume is calculated at 36 minutes after start, and estimated blood volume is computed 62 minutes after start.
  The primary outcome is the agreement between actual blood volume in ml (as measured via radiodilution by the BVA-100) and estimated blood volume (as measured the methods described in arm 2).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Wofford, PhD, Principal Investigator — Uniformed Services University of the Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Conzen P, Rehm M. A rational approach to perioperative fluid management. Anesthesiology. 2008 Oct;109(4):723-40. doi: 10.1097/ALN.0b013e3181863117. PMID 18813052
- [Background] D'Angelo MR, Dutton RP. Hemodynamic measurement in the operating room: a review of conventional measures to identify hypovolemia. AANA J. 2009 Aug;77(4):279-84. PMID 19731846
- [Background] Gallagher K, Vacchiano C. Reexamining traditional intraoperative fluid administration: evolving views in the age of goal-directed therapy. AANA J. 2014 Jun;82(3):235-42. PMID 25109164
- [Background] Johnson A, Ahrens T. Stroke volume optimization: the new hemodynamic algorithm. Crit Care Nurse. 2015 Feb;35(1):11-27. doi: 10.4037/ccn2015427. PMID 25639574
- [Background] Joosten A, Alexander B, Cannesson M. Defining goals of resuscitation in the critically ill patient. Crit Care Clin. 2015 Jan;31(1):113-32. doi: 10.1016/j.ccc.2014.08.006. PMID 25435481
- [Background] Peng K, Li J, Cheng H, Ji FH. Goal-directed fluid therapy based on stroke volume variations improves fluid management and gastrointestinal perfusion in patients undergoing major orthopedic surgery. Med Princ Pract. 2014;23(5):413-20. doi: 10.1159/000363573. Epub 2014 Jul 3. PMID 24994571
- [Background] Ramsingh DS, Sanghvi C, Gamboa J, Cannesson M, Applegate RL 2nd. Outcome impact of goal directed fluid therapy during high risk abdominal surgery in low to moderate risk patients: a randomized controlled trial. J Clin Monit Comput. 2013 Jun;27(3):249-57. doi: 10.1007/s10877-012-9422-5. Epub 2012 Dec 22. PMID 23264068
- [Background] Scheeren TW, Wiesenack C, Gerlach H, Marx G. Goal-directed intraoperative fluid therapy guided by stroke volume and its variation in high-risk surgical patients: a prospective randomized multicentre study. J Clin Monit Comput. 2013 Jun;27(3):225-33. doi: 10.1007/s10877-013-9461-6. Epub 2013 Apr 5. PMID 23558909
- [Background] Aya HD, Cecconi M, Hamilton M, Rhodes A. Goal-directed therapy in cardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):510-7. doi: 10.1093/bja/aet020. Epub 2013 Feb 27. PMID 23447502
- [Background] Correa-Gallego C, Tan KS, Arslan-Carlon V, Gonen M, Denis SC, Langdon-Embry L, Grant F, Kingham TP, DeMatteo RP, Allen PJ, D'Angelica MI, Jarnagin WR, Fischer M. Goal-Directed Fluid Therapy Using Stroke Volume Variation for Resuscitation after Low Central Venous Pressure-Assisted Liver Resection: A Randomized Clinical Trial. J Am Coll Surg. 2015 Aug;221(2):591-601. doi: 10.1016/j.jamcollsurg.2015.03.050. Epub 2015 Apr 7. PMID 26206652
- [Background] Van PY, Riha GM, Cho SD, Underwood SJ, Hamilton GJ, Anderson R, Ham LB, Schreiber MA. Blood volume analysis can distinguish true anemia from hemodilution in critically ill patients. J Trauma. 2011 Mar;70(3):646-51. doi: 10.1097/TA.0b013e31820d5f48. PMID 21610355
- [Background] Borovka M, Teruya S, Alvarez J, Helmke S, Maurer MS. Differences in blood volume components between hyporesponders and responders to erythropoietin alfa: the heart failure with preserved ejection fraction (HFPEF) anemia trial. J Card Fail. 2013 Oct;19(10):685-91. doi: 10.1016/j.cardfail.2013.08.508. PMID 24125107
- [Background] Feldschuh J, Enson Y. Prediction of the normal blood volume. Relation of blood volume to body habitus. Circulation. 1977 Oct;56(4 Pt 1):605-12. doi: 10.1161/01.cir.56.4.605. PMID 902387
- [Background] Feldschuh J, Katz S. The importance of correct norms in blood volume measurement. Am J Med Sci. 2007 Jul;334(1):41-6. doi: 10.1097/MAJ.0b013e318063c707. PMID 17630591
- [Background] D'Angelo M, Hodgen RK, Wofford K, Vacchiano C. A Theoretical Mathematical Model to Estimate Blood Volume in Clinical Practice. Biol Res Nurs. 2015 Oct;17(5):478-86. doi: 10.1177/1099800414555410. Epub 2014 Oct 20. PMID 25332464